CLINICAL TRIAL: NCT01586728
Title: Indication and Benefits of Nocturnal Oxygen Therapy in Cystic Fibrosis
Brief Title: Oxygen Therapy in Cystic Fibrosis
Acronym: MUCOXY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusion in the study
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P 100801
Record Dates: First submitted 2012-01-18; First posted 2012-04-27 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; oxygen therapy; sleep
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air - oxygen (Other): One period in room air and one period with nocturnal oxygen therapy, separated by a wash out period of 2 to 6 weeks.
  Interventions: Other: Air - oxygen
- Oxygen - Air (Other): One period with nocturnal oxygen therapy and one period in room air, separated by a wash out period of 2 to 6 weeks.
  Interventions: Other: Oxygen - Air

INTERVENTIONS:
Other: Air - oxygen — 1. his routine long term treatment without nocturnal oxygen therapy during 6 weeks (air period)
  2. nocturnal oxygen therapy with a stable flow to obtain a nocturnal SpO2 > 90% (oxygen period) while continuing his routine long term treatment during 6 weeks.
  During the oxygen period, the oxygen flow will be at least 1.5l/min. This flow may be increased up to 2L/min in case of the presence of nocturnal periods with SpO2 <= 90%.
  Arms: Air - oxygen
Other: Oxygen - Air — 1. nocturnal oxygen therapy with a stable flow to obtain a nocturnal SpO2 > 90% (oxygen period) while continuing his routine long term treatment during 6 weeks.
  2. his routine long term treatment without nocturnal oxygen therapy during 6 weeks (air period) During the oxygen period, the oxygen flow will be at least 1.5l/min. This flow may be increased up to 2L/min in case of the presence of nocturnal periods with SpO2 <= 90%.
  Arms: Oxygen - Air

SUMMARY:
This is an open, multicenter, prospective, randomised and cross over study, comparing in patients with cystic fibrosis aged > 6 years, 2 periods of 6 weeks of oxygen therapy or room air, separated by a wash out period of 2 to 6 weeks.

DETAILED DESCRIPTION:
Rationale Oxygen therapy may be proposed to patients with cystic fibrosis (CF) with nocturnal hypoxemia but the indication and benefits of oxygen therapy have not been validated in CF.

Aim of the study and main objective The aim of the study is to evaluate the improvement in nocturnal hypoxemia by the measurement of nocturnal pulse oximetry (SpO2) after 6 weeks of nocturnal oxygen therapy in stable patients with CF.

An improvement is defined by a nocturnal SpO2 > 90% during the whole night.

Objectives and secondary aims

* Comparison of subjective sleep quality during oxygen therapy and room air after a period of 6 weeks by means of 4 validated sleep questionnaires
* Comparison of quality of life during oxygen therapy and room air after a period of 6 weeks by means of a validated questionnaire for CF patients (CFQ).
* Detection of the appearance or increase in nocturnal hypercapnia during oxygen therapy and room air after a period of 6 weeks
* Comparison of a possible arterial pulmonary hypertension during oxygen therapy and room air after a period of 6 weeks by means of an echocardiography

Study design This is an open, multicentre, prospective, randomised and cross over study, comparing in individual patient two periods of 6 weeks: one period with nocturnal oxygen therapy and one period in room air, separated by a wash out period of 2 to 6 weeks.

Inclusion criteria

* Children ≥ 6 years and adults ≥ 18 years with CF in a stable state
* With a forced expiratory volume in one second (FEV1) ≤ 50% of predicted value
* Having a pulse oximetry (SpO2) in room air ≤ 90% for ≥ 10% of the night and/or a SpO2 ≤ 90% for ≥ 10 minutes during the night
* Any patient with prior noninvasive positive pressure ventilation (NPPV) but who has stopped NPPV at least 15 days before the start of the study.
* Written approval by the patient and by the parents in case of a pediatric patient
* Patient having the French social security coverage Non-inclusion criteria
* Patients with a respiratory exacerbation during the last 15 days
* Patients with NPPV or long term oxygen therapy prior to the start of the study and unable to stop this treatment
* Impossibility of a medical examination
* Pregnant patient or breastfeeding patient

Study protocol The study is proposed to the patients during the V0 visit, corresponding to the screening monitoring showing a nocturnal SpO2 in room air ≤ 90% for ≥ 10% of the night and/or a SpO2 ≤ 90% for ≥ 10 minutes during the night. After a period of 2 to 30 days, the written approval is obtained during a routine visit.

Thereafter, the patient will be randomised to receive either:

1. nocturnal oxygen therapy with a stable flow to obtain a nocturnal SpO2 >90% (Oxygen period) while continuing his routine long term treatment
2. his routine long term treatment without nocturnal oxygen therapy (Air period) During the Oxygen period, the oxygen flow will be at least 1.5 L/min. This flow may be increased up to 2L/min in case of the presence of nocturnal periods with a SpO2 ≤ 90%.

The two periods Oxygen and Air will be separated by a wash out period of 2 to 6 weeks to rule out any long lasting effect of nocturnal oxygen therapy.

At the end of the 2 periods of 6 weeks oxygen or air, the following investigations will be performed:

* A nocturnal evaluation of gas exchange by the Sentec™ monitor (which measures SpO2 and transcutaneous carbon dioxide (PCO2)) and objective sleep quality by means of actigraphy
* an evaluation of subjective sleep quality by means of 4 validates sleep questionnaires
* an evaluation of quality of life by a validated CF questionnaire (CFQ)
* spirometry with blood gases in room air
* an echocardiography

Number of subjects Only 3 studies have evaluated the benefit of oxygen therapy on nocturnal gas exchange during one night and only one study has evaluated the benefit of oxygen therapy after a period of 26 months. This last study is limited by the small number of patients and the low compliance with oxygen therapy.

No study has evaluated the effect of oxygen therapy during a 6 weeks period. This limits the calculation of the number of subjects.

As the study is a cross over study, a number of 30 analysable patients is estimated to be sufficient for the evaluation of the primary outcome measure and the secondary outcomes. Because of the possibility of premature withdrawal, it is planned to include 50 patients.

Total duration of the study: maximum 22.5 months

Inclusion period: 18 months

Duration of participation for one patient: maximum 4.5 months

Statistical analysis and final report: 3 months

Number of participating centres: 8

Estimation of the mean number of patients included per centre: 3 patients / 3 months / centre

Expected results The results of the present study should help to define the criteria to start long term oxygen therapy and to assess the potential benefits of this treatment in stable patients with CF.

ELIGIBILITY:
Inclusion Criteria:

* Children ≥ 6 years and adults ≥ 18 years with CF in a stable state
* With a forced expiratory volume in one second (FEV1) ≤ 50% of predicted value
* Having a pulse oximetry (SpO2) in room air ≤ 90% for ≥ 10% of the night and/or a SpO2 ≤ 90% for ≥ 10 minutes during the night
* Any patient with prior noninvasive positive pressure ventilation (NPPV) but who has stopped NPPV at least 15 days before the start of the study.
* Written approval by the patient and by the parents in case of a pediatric patient
* Patient having the French social security coverage

Exclusion Criteria:

* Patients with a respiratory exacerbation during the last 15 days
* Patients with NPPV or long term oxygen therapy prior to the start of the study and unable to stop this treatment
* Impossibility of a medical examination
* Pregnant patient or breastfeeding patient

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
the improvement in nocturnal hypoxemia by the measurement of nocturnal pulse oximetry (SpO2) after 6 weeks of nocturnal oxygen therapy in stable patients with CF | after a 6 weeks period

SECONDARY OUTCOMES:
Comparison of subjective sleep quality during oxygen therapy and room air after a period of 6 weeks by means of 4 validated sleep questionnaires | after a 6 weeks period
Comparison of quality of life during oxygen therapy and room air after a period of 6 weeks by means of a validated questionnaire for CF patients (CFQ). | after a 6 weeks period
Detection of the appearance or increase in nocturnal hypercapnia during oxygen therapy and room air after a period of 6 weeks | after a 6 weeks period
Comparison of a possible arterial pulmonary hypertension during oxygen therapy and room air after a period of 6 weeks by means of an echocardiography | after a 6 weeks period

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte FAUROUX, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de pneumologie pédiatrique, Hôpital Armand Trousseau, Paris, France